CLINICAL TRIAL: NCT03579446
Title: Levorphanol as a Second Line Opioid in Cancer Patients Undergoing Opioid Rotation: An Open Label Study
Brief Title: Levorphanol as a Second Line Opioid in Reducing Pain in Patients With Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: <75% participation
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-0925; NCI-2018-01139 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0925 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasm Metastasis | interventions — Hydrocodone; Hydromorphone; Levorphanol; Morphine; Oxycodone; Oxymorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supportive care (levorphanol, opioid regimen) (Experimental): Patients receive levorphanol PO every 8 or 12 hours for 30 days. Patients may receive opioid regimen including hydrocodone, morphine, hydromorphone, oxycodone, and oxymorphone for breakthrough pain. Patients may continue levorphanol for an additional 6-8 months if it is determined by the Principal Investigator the patient can continue.
  Interventions: Drug: Hydrocodone; Drug: Hydromorphone; Drug: Levorphanol; Drug: Morphine; Drug: Oxycodone; Drug: Oxymorphone; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Hydrocodone — Given by PO
Drug: Hydromorphone — Given by PO
  Other Names: (-)-Hydromorphone; Dihydromorphinone; Hydromorphon
Drug: Levorphanol — Given PO
Drug: Morphine — Given by PO
Drug: Oxycodone — Given by PO
  Other Names: Oxycodone SR
Drug: Oxymorphone — Given by PO
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This early phase I trial studies how well levorphanol works as a second line opioid in reducing pain in patients with cancer that may have spread to other places in the body. Levorphanol may work better in controlling cancer pain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the proportion of successful opioid rotation (OR) from morphine equivalent daily dose (MEDD) to levorphanol at the primary end point.

SECONDARY OBJECTIVES:

I. To determine the median opioid rotation ratio (ORR) in patients undergoing successful opioid rotations from morphine equivalent daily dose (MEDD) to levorphanol in the Supportive Care Center (SCC) or Pain Clinic.

II. To determine the effect of levorphanol on cancer pain (as measured by change in Edmonton Symptom Assessment System's [ESAS] pain item from baseline) in cancer outpatients undergoing opioid rotation to levorphanol at the primary end point of treatment.

III. To determine the association between the opioid rotation ratio from MEDD to levorphanol and baseline MEDD prior to opioid rotation.

IV. Measure levorphanol related side effects using the opioid side effect scale at day 10 +/- 1 of starting levorphanol.

V. Determine what percentage of patients rotated to levorphanol achieve their personalized pain goal.

VI. Determine the predictors of successful opioid rotation from other opioids to levorphanol.

OUTLINE:

Patients receive levorphanol orally (PO) every 8 or 12 hours for 30 days. Patients may receive opioid regimen including hydrocodone, morphine, hydromorphone, oxycodone, and oxymorphone for breakthrough pain. Patients may continue levorphanol for an additional 6-8 months if it is determined by the Principal Investigator the patient can continue.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen in the SCC or Pain Clinic with a diagnosis of cancer with or without evidence of metastatic disease
* Diagnosis of cancer related pain currently treated with first line strong oral opioid analgesics such as morphine, oxycodone, oxymorphone, hydromorphone or hydrocodone
* Age 18 or older
* Able to complete study assessments
* Individual is willing to sign written informed consent
* Patients who are classified as being opioid tolerant by receiving a baseline MEDD of >= 60 mg
* Patients who are local and able to follow-up in the SCC or Pain Clinic within 30 days if necessary
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 3

Exclusion Criteria:

* Cognitive impairment with a Memorial Delirium Assessment Scale (MDAS) score of 7 or higher or diagnosed with neurocognitive impairment by the treating SCC or Pain Clinic physician
* Renal insufficiency defined as estimated glomerular filtration rate of < 60
* Hepatic insufficiency defined as transaminitis (aspartate aminotransferase [AST] or alanine aminotransferase [ALT] > 3 times the highest normal value) or hyperbilirubinemia of > 1.5 times the highest normal value
* Non-English speaking participants as not all assessments are validated in other languages
* Presence of neuropathic pain as a primary pain syndrome
* Non-malignant pain
* Patients with history of alcohol or substance abuse by using Cut-down, Annoyed, Guilty, Eye-opener adapted to include Drug use questionnaire (CAGE-AID) score of 2 or higher; Pain Clinic: Screener and Opioid Assessment for Patients with Pain (SOAPP) score of 7 or higher. In the unlikely event that CAGE-AID or SOAPP is not present in patient's chart, a CAGE-AID questionnaire will be administered after obtaining verbal consent for screening
* Patients receiving methadone due to reasons such as long and variable half-life
* Patients receiving scheduled benzodiazepines due to the risk of excessive sedation
* Patients with a MEDD of > 300
* Unable or unwilling to sign consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Proportion of successful opioid rotation (OR) from morphine equivalent daily dose (MEDD) to levorphanol | Day 10 or any day after 2 days of rotation to levorphanol
  Bayesian methodology developed by Peter Thall will be used to monitor the study. This method decides whether levorphanol is promising relative to the standard medicine. Will estimate the proportion of successful opioid rotation along with a 95% confidence interval. Association between successful opioid rotation and demographic/clinical characteristics will be examined by Chi-squared test or Fisher's exact test when appropriate. Logistic regression model will be employed to assess the effect of demographic/clinical characteristics on the presence of successful opioid rotation.

SECONDARY OUTCOMES:
Opioid rotation ratio (ORR) | Up to 30 days
  Will be calculated by levorphanol mg (day 10 +/- 1) over MEDD (day 0). ORR will be summarized using standard descriptive statistics such as mean, standard deviation, median and range. Wilcoxon rank-sum test or Kruskal-Wallis test will be applied to examine the difference on ORR between/among patients' characteristics groups.
Change of Edmonton Symptom Assessment Scale (ESAS) pain score | Baseline up to day 10 or any day after 2 days of rotation to levorphanol
  Pain score change will be summarized using standard descriptive statistics such as mean, standard deviation, median and range. Wilcoxon rank-sum test or Kruskal-Wallis test will be applied to examine the difference on pain score change between/among patients' characteristics groups. Since ESAS pain score will be measured daily from day 0 to day 10 +/- 1 and on day 30 +/- 3, mixed model will be applied to examine the differential changes over time for ESAS pain score, adjusting for other covariates of interest. ORR and baseline MEDD will be presented by scatter plots. Correlation will be assessed between levorphanol dose on day 10 +/- 1, ORR and baseline MEDD suing Pearson or Spearman correlation coefficient when appropriate. Linear regression models will be applied to estimate the linear association between levorphanoal dose on day 10 +/- 1, ORR and baseline MEDD.
Incidence of levorphanol related side effects | Up to day 30
  Will be rated using the Opioid Side Effect Scale on xerostmia, nauseas, constipation, drowsiness and confusion daily from day 0 to day 10 +/-1 and on day 30 +/- 3.
Personalized pain goal (PPG) | Up to day 30
  PPG will be summarized using standard descriptive statistics such as mean, standard deviation, median and range. Mixed model will be applied to examine the differential changes over time for opioid side effect scale, adjusting for other covariates of interest. The goal is not achieved if the PPG is lower than the ESAS pain score. Frequency and proportion of achieved goal will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Akhila S Reddy, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2020-01-02): https://cdn.clinicaltrials.gov/large-docs/46/NCT03579446/ICF_000.pdf